CLINICAL TRIAL: NCT03457038
Title: Use of Fc Mannose-Binding Lectin to Detect and Monitor the Presence of Pathogen-Associated Molecular Patterns During Septic Shock
Brief Title: Use of Fc-MBL to Detect and Monitor the Presence of PAMPs During Septic Shock
Acronym: Fc-MBL/PAMPs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0157; 2017-A01686-47 (Other: ID-RCB)
Record Dates: First submitted 2018-02-26; First posted 2018-03-07 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Septic Shock
Keywords: Mannose-Binding Lectin, PAMPs,
MeSH Terms: conditions — Shock, Septic | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Major patients admitted to the Resuscitation Department of the CHU Toulouse-Rangueil for severe sepsis, or development of sepsis during the stay resuscitation; sepsis defined by a SOFA score ≥ 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Septic Shock (Experimental): Patient Hospitalized in Intensive Care Unit for sepsis of any etiology. The number of follow-up visits will not be changed compared to usual patient follow-up hospitalized in the intensive care unit but there will be blood testing more frequently
  Interventions: Biological: Blood Test

INTERVENTIONS:
Biological: Blood Test — Addition to the current care but during the normal follow-up visit :
  * At the entrance to the service: search for bacterial 16S RNA in the blood
  * Additional blood tests (4) at T6-12-18 and 36h
  * At each visit: Sampling of an additional heparinized blood tube for the assay PAMPs.
  * 1 time per day: Assay of CRP and PCT from samples taken in common practice
  * J30: Assessment of the vital status of the patient

SUMMARY:
Use Mannose Binding Lectin (MBL) as a biomarker to measure levels of Pathogen- Associated Molecular Patterns (PAMP) during septic shock. This will allow evaluating interest of this biomarker to monitor and manage a septic shock. Consecutive patients admitted for sepsis in Intensive Care Unit Department will be included. This biomarker will be compared to all the parameters monitored usually for these patients in standard care.

DETAILED DESCRIPTION:
Septic shock still represent a major cause of admission in intensive care unit, incidence of severe sepsis is increasing, even in western countries, due to aging populations and comorbidities. Definition of septic shock was revised in 2016 by a task force, which emphasizes the need for future iterations. Indeed, there are no simple clinical or biological criteria ton diagnose septic patients with high risk of shock, or to prognose its severity. C-reactive protein (CRP) and procalcitonin (PCT) are the wider biomarkers used to monitor septic patients. But they do not correlate with sepsis severity and moreover do not distinguish unequivocally between infection and noninfected systemic inflammatory response syndrome (SIRS). Each microorganism has number of PAMPs, cell wall components (lipopolysaccharide endotoxin, peptidoglycan, outer membrane vesicles), flagella, mannan… High levels of these pathogen fragments are released in the bloodstream during sepsis. They trigger release of inflammatory cytokines that drive the sepsis cascade. Mannose binding lectin plays a pivotal role in innate immunity, binding with surface sugars of wide range of pathogens and their fragments. Thus MBL promotes opsonophagocytosis and activates the lectin-complement pathway. Fc-MBL, an engineered version of MBL has been developed to capture microorganism and treat sepsis. An ELISA, using Fc-MBL was developed to measure PAMPs in whole blood during sepsis. This assay will use Fc-MBL ELISA to quantify PAMPs during septic shock, to improve diagnostic and monitoring. But also, identifying patients with high levels of PAMPs for dialysis-like sepsis therapies.

PAMP's level will be compared to clinical, biological, microbiological and therapeutic outcomes. Its sensitivity will be evaluated by its kinetic among a septic shock (defined with Sepsis-3 criteria) and by correlation with CRP (C-Reactive Protein) and PCT (Procalcitonin). Its specificity will be evaluated by comparing its levels during septic and non-septic shocks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Hospitalized in Intensive Care Unit for sepsis of any etiology
* Patients with shock criteria: defined by a hypotension, hyperlactatemia, the use of vasopressive drugs.
* Patient affiliated to a social security scheme- Patient giving consent

Exclusion Criteria:

* Minor patients
* Organ transplant
* Immunosuppressive drugs, other than corticosteroids
* Patients who decline participating to the assay
* Persons placed under legal protection, guardianship
* Pregnant woman
* Subject participating in another search including a exclusion period still in progress at pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-07-18 (Estimated); Study Completion 2019-07-18 (Estimated)

PRIMARY OUTCOMES:
Quantify in whole blood presence of PAMP during a septic shock, | Follow-up during 30 days
  Quantify in whole blood presence of PAMP during a septic shock, using Fc-MBL ELISA :t o improve diagnostic by distinguishing a septic shock from another shock, and stating prognosis by studying PAMP kinetic under antibiotherapy.

SECONDARY OUTCOMES:
Compare accuracy of Fc-MBL ELISA PAMP assay to CRP and PCT during septic shock. | Follow-up during 30 days
  PAMP's level will be compared to clinical, biological, microbiological and therapeutic outcomes. Its sensitivity will be evaluated by its kinetic among a septic shock (defined with Sepsis-3 criteria) and by correlation with CRP and PCT. Its specificity will be evaluated by comparing its levels during septic and non-septic shocks.
Study PAMP's kinetic during septic shock from various origins | Follow-up during 30 days
  PAMP's level will be compared to clinical, biological, microbiological and therapeutic outcomes. Its sensitivity will be evaluated by its kinetic among a septic shock (defined with Sepsis-3 criteria) and by correlation with CRP and PCT. Its specificity will be evaluated by comparing its levels during septic and non-septic shocks.
Identify patients who could beneficiate to a dialysis-like therapy | Follow-up during 30 days
  identifying patients with high levels of PAMPs for dialysis-like sepsis therapies

CONTACTS AND LOCATIONS:
Overall Officials: Eric Oswald, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bicart-See A, Vardon F, Ruiz S, Conil JM, Tudal V, Super M, Ingber DE, Oswald E. Kinetics of molecular patterns captured by mannose-binding lectin in septic shock correlate with clinical outcome: a monocentric prospective observational study. Intensive Care Med Exp. 2025 Dec 10;13(1):123. doi: 10.1186/s40635-025-00832-x. PMID 41366523